CLINICAL TRIAL: NCT06295120
Title: The Optimal Antibiotic Treatment Duration for Community-acquired Pneumonia in Adults Diagnosed in General Practice in Denmark: an Open-Label, Pragmatic, Randomised Controlled Trial
Brief Title: The Optimal Antibiotic Treatment Duration for Community-acquired Pneumonia in Adults Diagnosed in General Practice in Denmark (CAP-D)
Acronym: CAP-D
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Research Unit for General Practice in Aalborg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 362-1
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-11

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-acquired pneumonia; Treatment duration; Phenoxymethylpenicillin; General Practice
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 3 days (Experimental): 3 days of treatment with phenoxymethylpenicillin 1.2 MIE 4 times daily.
  Interventions: Drug: Phenoxymethylpenicillin 1.2 MIE 4 times daily
- 4 days (Experimental): 4 days of treatment with phenoxymethylpenicillin 1.2 MIE 4 times daily.
  Interventions: Drug: Phenoxymethylpenicillin 1.2 MIE 4 times daily
- 5 days (Experimental): 5 days of treatment with phenoxymethylpenicillin 1.2 MIE 4 times daily.
  Interventions: Drug: Phenoxymethylpenicillin 1.2 MIE 4 times daily
- 6 days (Experimental): 6 days of treatment with phenoxymethylpenicillin 1.2 MIE 4 times daily.
  Interventions: Drug: Phenoxymethylpenicillin 1.2 MIE 4 times daily
- 7 days (Active Comparator): 7 days of treatment with phenoxymethylpenicillin 1.2 MIE 4 times daily.
  Interventions: Drug: Phenoxymethylpenicillin 1.2 MIE 4 times daily

INTERVENTIONS:
Drug: Phenoxymethylpenicillin 1.2 MIE 4 times daily — The intervention is the duration of treatment with phenoxymethylpenicillin from 3 to 7 days. Dose and frequency of the treatment is the same in the different arms.

SUMMARY:
The aim of this randomised controlled trial is to identify the optimal treatment duration with phenoxymethylpenicillin for community-acquired pneumonia diagnosed in general practice.

Eligible participants are adults (≥18 years) presenting in general practice with symptoms of an acute LRTI (i.e., acute illness (≤ 21 days) usually with cough and minimum one other symptom such as dyspnea, sputum production, wheezing, chest discomfort or fever) in whom the GP finds it relevant to treat with antibiotics.

Consenting patients who meet all the eligibility criteria will be randomised (1:1:1:1:1) to either three, four, five, six or seven days of treatment with phenoxymethylpenicillin 1.2 MIE four times daily.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants are adults (≥18 years) presenting in general practice with symptoms of an acute LRTI (i.e., acute illness (≤ 21 days) usually with cough and minimum one other symptom such as dyspnoea, sputum production, wheezing, chest discomfort or fever) in whom the GP finds it relevant to treat with antibiotics.

Exclusion Criteria:

1. Need for immediate hospitalisation at the time of diagnosis.
2. Known allergy to beta-lactam antibiotics.
3. Any coinfection necessitating antibiotic treatment.
4. Use of systemic antibiotics or antivirals within the last month.
5. Pre-existing lung disease (e.g., chronic obstructive pulmonary disease, bronchiectasis, asthma, lung cancer).
6. Known immunosuppression (i.e., long term treatment with corticosteroid, chemotherapy, or immune disorder).
7. Pregnant or lactating.
8. Patients not capable of consenting and/or patients deemed non-suitable for participation by the healthcare professional.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment failure at day 30 | From randomisation to day 30
  Treatment failure is defined as any hospitalisation OR change in the antibiotic strategy (i.e., prolongation of the duration, change in antibiotic type, new antibiotic prescription) due to symptoms of acute respiratory tract infection - between randomisation and day 30.

SECONDARY OUTCOMES:
Clinical recovery at day 8 | From randomisation to day 8
  Clinical recovery is defined as: The participant scores below a pre-defined cut-off point for being recovered at the Acute Respiratory Tract Infection Questionnaire OR reports feeling recovered by themselves AND the participant is no longer treated with any antibiotics.
The Acute Respiratory Tract Infection Questionnaire (ARTIQ) score | At randomisation day and day 8
  The Acute Respiratory Tract Infection Questionnaire is a validated, self-administered, multidimensional, sum-scaling symptom score monitoring the severity and functional impact of acute respiratory tract infections in general practice. The questionnaire consists of five single items and 37 items covering five independent dimensions: upper respiratory tract symptoms, lower respiratory tract symptoms, physiological, sleep, and medicine. The participants will be asked to evaluate each item, over the past 24 hours by using a three-point scale: "No (0 point)", "Yes - some (1 point)" or "Yes - a lot (2 points)". Ten items are dichotomized: "Yes (1 point) or "No (0 point)"). The total ARTIQ score is calculated as the sum of each dimension and single items (minimum 0 - maximum 74).
Prolonged antibiotic treatment | From randomisation to day 30
  Proportion of participants in need of prolonged antibiotic treatment.
Change in type of antibiotic | From randomisation to day 30
  Proportion of participants who had prescribed another type of antibiotic treatment
Relapse of acute Lower Respiratory Tract Infection (LRTI) | From randomisation to day 30
  Proportion of participants with relapse of acute LRTI
Reconsultation | From randomisation to day 30
  Number of reconsultations at general practice or out-off-hour services
New prescriptions within 30 days | From randomisation to day 30
  Proportion of participants with new prescriptions of symptomatic treatment (e.g. prednisolone, bronchodilator etc) within 30 days
Hospitalisation | From randomisation to day 30
  Proportion of participants hospitalised within 30 days
Mortality | From randomisation to day 30
  All-cause mortality at day 30
Adverse events | From randomisation to day 30
  Proportion of participants experiencing adverse or serious adverse events
Treatment adherence | From randomisation to day 8
  Initiation, implementation and discontinuation of the allocated treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Research Unit for General Practice Aalborg, Gistrup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johansen E, Nielsen H, Gillespie D, Aabenhus R, Hansen MP. The optimal antibiotic treatment duration for community-acquired pneumonia in adults diagnosed in general practice in Denmark (CAP-D): an open-label, pragmatic, randomised controlled trial. Trials. 2024 Sep 27;25(1):627. doi: 10.1186/s13063-024-08477-z. PMID 39334468